CLINICAL TRIAL: NCT01295372
Title: A 6-month, Randomised, Double-blind, Parallel-group, Risperidone-controlled, Fixed-dose Study Evaluating the Safety and Efficacy of Zicronapine in Patients With Schizophrenia
Brief Title: Safety and Efficacy of Zicronapine in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13639A; 2010-022181-28 (EudraCT Number)
Record Dates: First submitted 2011-02-03; First posted 2011-02-14 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Antipsychotic; Risperidone; Lu 31-130
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zicronapine (Experimental)
  Interventions: Drug: Zicronapine
- Risperidone (Active Comparator)
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Zicronapine — 7.5 mg/day; orally
  Other Names: Past name: Lu 31-130
  Arms: Zicronapine
Drug: Risperidone — 5 mg/day; orally
  Other Names: Risperdal®
  Arms: Risperidone

SUMMARY:
To assess the effect of zicronapine versus risperidone on metabolic parameters comprising body weight, body mass index (BMI), waist circumference, levels of fasting blood lipids and glucose during 6 months of treatment.

DETAILED DESCRIPTION:
Schizophrenia is a serious and disabling mental disorder that affects approximately 1% of the world's population. Antipsychotic drugs remain the cornerstone in the pharmacotherapy of schizophrenia. There are a number of antipsychotic drugs in use but none is ideal, in particular because their safety profile is complex and their effectiveness is limited.

Thus, present treatment options leave room for improvement and call for new, more effective pharmacotherapies for the treatment of schizophrenia. In the current study, non-acute patients with schizophrenia will be randomised to blinded treatment with either zicronapine or a standard antipsychotic treatment for 24 weeks. The safety (with focus on metabolic parameters) and efficacy of zicronapine will be evaluated in comparison to risperidone.

ELIGIBILITY:
Inclusion Criteria:

* The patient meets the Diagnostic and Statistical Manual of Mental Disorders, 4th edition, Text Revision (DSM-IV-TR) criteria for schizophrenia
* The patient is a man or woman, ≥18 and ≤65 years old
* The patient has a PANSS total score ≥60 and ≤100 (extremes included) at screening and baseline

Exclusion Criteria:

* The patient has a current, predominant Axis I psychiatric disorder other than schizophrenia as defined in the DSM-IV-TR
* The patient has a current diagnosis or a history of substance dependence (except nicotine) or substance abuse (except cannabis) according to the DSM-IV-TR criteria ≤6 months prior to screening
* The patient is at significant risk of harming him/herself or others according to the investigator's judgement (assisted by the assessment of suicidal ideation and behaviour using the C-SSRS)
* The patient is resistant to antipsychotic treatment according to the investigator's judgement or has been treated with clozapine ≤3 months prior to screening
* The patient has experienced an acute exacerbation requiring hospitalisation ≤3 months prior to screening or between screening and baseline
* The patient has been treated with risperidone or paliperidone ≤6 months prior to screening

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2011-04; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To assess the effect of zicronapine versus risperidone on body weight (and BMI) | 6 months
To assess the effect of zicronapine versus risperidone on waist circumference | 6 months
To assess the effect of zicronapine versus risperidone on levels of fasting blood lipids | 6 months
To assess the effect of zicronapine versus risperidone on levels of fasting blood glucose | 6 months

SECONDARY OUTCOMES:
To assess the overall safety and tolerability of zicronapine versus risperidone during 6 months of treatment by comparing the frequencies of adverse events sorted by system organ class and preferred term. | 6 months
To assess the potential of zicronapine versus risperidone to induce extrapyramidal symptoms using change from baseline to each assessment in the AIMS, BARS, and SAS total scores | 6 months
  Abnormal Involuntary Movement Scale (AIMS), Barnes Akathisia Scale (BARS), and Simpson Angus Scale (SAS) total scores
To assess the effect of zicronapine versus risperidone on serum prolactin levels | 6 months
To assess the effect of zicronapine on suicidal ideation and behaviour using the Columbia Suicide-Severity Rating Scale (C-SSRS) | 6 months
To assess the effect of zicronapine versus risperidone on electrocardiogram (ECG) parameters | 6 months
To assess the efficacy of zicronapine versus risperidone following 6 months of treatment using change from baseline in the Positive and Negative Syndrome Scale (PANSS) total score | 6 months
To assess the efficacy of zicronapine versus risperidone using change from baseline to each assessment in the PANSS total score and PANSS subscale scores (Positive Symptoms, Negative Symptoms, and General Psychopathology) | 6 months
To assess the efficacy of zicronapine versus risperidone by comparing the proportions of responders (using two definitions of response: ≥20% and ≥50% decrease from baseline in PANSS total score) | 6 months
To assess the efficacy of zicronapine versus risperidone on global improvement using change from baseline to each assessment in the Clinical Global Impression - Severity of Illness (CGI-S) score | 6 months
To assess the effect of zicronapine versus risperidone on personal and social functioning using the Personal and Social Performance Scale (PSP) | 6 months
To assess the effect of zicronapine versus risperidone on functioning using the Global Assessment of Functioning scale (GAF) | 6 months
To assess the effect of zicronapine versus risperidone on quality of life using the disease-specific Schizophrenia Quality of Life scale (S-QoL) | 6 months
To assess the effect of zicronapine versus risperidone on the patient's satisfaction with treatment using the Medication Satisfaction Questionnaire (MSQ) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (24):
- Czechia (8):
  - CZ004, Brno
  - CZ001, Brno
  - CZ007, Kladno
  - CZ003, Liberec
  - CZ002, Olomouc
  - CZ008, Prague
  - CZ006, Prague
  - CZ005, Sternberk
- Estonia (4):
  - EE003, Pärnu
  - EE001, Tallinn
  - EE002, Tallinn
  - EE004, Tartu
- Finland (2):
  - FI001, Helsinki
  - FI002, Kellokoski
- France (4):
  - FR001, Clermont-Ferrand
  - FR002, Nîmes
  - FR004, Strasbourg
  - FR003, Toulon
- Poland (6):
  - PL004, Bełchatów
  - PL002, Gdansk
  - PL003, Kielce
  - PL006, Lodz
  - PL001, Lublin
  - PL005, Żuromin

REFERENCES:
- Available data/document: EudraCT Results: 2010-022181-28 — https://www.clinicaltrialsregister.eu/ctr-search/trial/2010-022181-28/result